CLINICAL TRIAL: NCT03325868
Title: Effect of Ulipristal Acetate on Bleeding Patterns and Dysmenorrhea in Women With Adenomyosis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: IND issues
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Cynthia Arvizo, Clinical Instructor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ulipristal
Record Dates: First submitted 2017-10-25; First posted 2017-10-30 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Adenomyosis; Heavy Uterine Bleeding; Dysmenorrhea
Keywords: heavy periods, painful periods, adenomyosis
MeSH Terms: conditions — Adenomyosis; Dysmenorrhea; Menorrhagia | interventions — ulipristal acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ulipristal (Experimental): Ulipristal acetate 5mg daily for 12 weeks
  Interventions: Drug: Ulipristal Acetate

INTERVENTIONS:
Drug: Ulipristal Acetate — Ulipristal 5mg daily by mouth for 12 weeks
  Other Names: Fibristal

SUMMARY:
Adenomyosis affects approximately 21% of symptomatic women who present to gynecology clinics. The disease is characterized by heavy bleeding and pain during periods. Limited treatment options exist for the treatment of adenomyosis for women who desire future child-bearing or prefer to avoid surgery. Recently, ulipristal acetate has been studied as a treatment option for women who have fibroids and heavy bleeding. The majority of women treated with ulipristal stopped having periods altogether. Our study aims to determine whether ulipristal is an adequate treatment for women with adenomyosis.

DETAILED DESCRIPTION:
Adenomyosis affects an estimated 20.9% of symptomatic women who present to gynecology clinics, with peak prevalence of 32% in 40-49 years old. Prior histologic studies in women undergoing hysterectomy show prevalence of with some variation due to differing histologic diagnostic criteria 10-37.1%. Heavy menstrual bleeding and dysmenorrhea are commonly manifested in women with adenomyosis. However, data on treatment of adenomyosis remains scarce. For women desiring definitive options, hysterectomy remains the treatment of choice. However, for women who desire future fertility, the currently accepted first-line therapy is progestogen therapy, particularly the levonorgestrel-IUD. Other limited studies have used danazol and GnRH agonists, but its use is limited by significant side effects.

Recently, the selective progesterone receptor modulators (SPRM) have emerged as successful medical treatment options for leiomyoma. The SPRM ulipristal acetate has been studied extensively in the treatment of leiomyoma and more recently endometriosis. Ulipristal acetate exerts both antagonist and agonist properties. Amenorrhea was achieved in 80% of women taking 5mg of ulipristal daily by treatment month 2 and up to 90% of women taking 10mg daily. Anovulation was achieved in 80% of women taking 5mg and 10mg dosing. Ulipristal acetate has not been studied as a treatment option for women with adenomyosis. We aim to study the effect of daily ulipristal on heavy menstrual bleeding in women with adenomyosis.

ELIGIBILITY:
Inclusion Criteria

* 18-51 years old
* PBAC score greater than 100
* Ultrasound or MRI findings of adenomyosis

Exclusion Criteria

* Inability to comprehend written and/or spoken English or Spanish
* Inability to provide informed consent
* Current uterine, breast, cervical or ovarian cancer
* Unwilling to use contraception
* Positive pregnancy test or planning pregnancy during the study period
* Submucosal uterine fibroids (or greater than a certain size)
* Current premalignancy or malignancy
* Endometrial ablation or uterine artery embolization
* Known hemoglobinopathy
* Known severe coagulation disorder
* Large uterine polyp (>2cm)
* BMI >40
* Previous or current treatment with SPRM or GnRH agonist
* Progestins, acetylsalicylic acid, mefenamic acid, anticoagulants, antifibrinolytic drugs, systemic glucocorticoids within 1 month of enrollment

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 0 (Actual)
Dates: Start 2018-02 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Bleeding patterns | 6 months
  Patient will use the pictorial blood loss assessment chart (PBAC) to describe bleeding patterns

SECONDARY OUTCOMES:
Quality of life | 6 months
  Patient will complete menorrhagia impact questionnaire (0-100, 0 is worst and 100 is best quality of life)
Pain | 6 months
  Patient will complete pain scale (0-10, 0 is no pain and 10 is worst pain)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Yunker, DO, Study Director — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No